CLINICAL TRIAL: NCT02259738
Title: Multi-modality MRI Study on Effect to Collateral Circulation and Blood Perfusion of Acute Cerebral Infarction by Human Urinary Kallidinogenase
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XuanwuH 2 (Other)
Responsible Party: Sponsor-Investigator, XuanwuH 2, Chief physician, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: hanying1
Record Dates: First submitted 2014-09-16; First posted 2014-10-08 (Estimated); Last update posted 2014-10-08 (Estimated); Status verified 2014-10

CONDITIONS: Cerebral Infarction
MeSH Terms: conditions — Cerebral Infarction | interventions — shuxuening

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human urinary kallidinogenase and Shuxuening injection (Experimental): Human urinary kallidinogenase 0.15PNA and Shuxuening injection 20mg, every day for 7 days.
  Interventions: Drug: Human Urinary Kallidinogenase; Drug: Shuxuening injection

INTERVENTIONS:
Drug: Human Urinary Kallidinogenase
  Other Names: youruikelin
Drug: Shuxuening injection

SUMMARY:
Human urinary kallidinogenase can promote the establishment of collateral circulation in the ischemic penumbra due to the stenosis or occlusion of middle cerebral artery and then increase the perfusion.

DETAILED DESCRIPTION:
Patients with acute ischemic stroke will be given human urinary kallidinogenase .Then we will estimate the cerebral collateral circulation in ischemic regions and final infarct volume, comparing with traditional therapy such as Shuxuening injection, which will provide new evidence for the treatment of ischemic stroke. Perfusion Weighted Imaging(PWI) could be a method to reflect the infarction center and low perfusion of tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age:greater than or equal to 18 years old and less than or equal to 70 years old;
* Time of onset is less than 7 days;
* Acute cerebral infarction due to the stenosis or occlusion of middle cerebral artery diagnosed by CT or MRI;
* The National Institute of Health Stroke Scale(NIHSS) score is 4 to 20;
* Excluding intracranial hemorrhage using CT or MRI.

Exclusion Criteria:

* The NIHSS score is less than or equal to 3;
* Patients with cerebral aneurysm, cerebral hemorrhage, brain tumor, brain contusion and laceration of brain and other diseases;
* Intracranial hemorrhage displaying by CT or MRI; Cardiac insufficiency;
* Cardiac insufficiency;
* Chronic liver disease(A/G inversion),elevated alanine aminotransferase(ALT)(more than 1.5 times the normal value);
* Increased serum creatinine(more than 1.5 times the normal value);
* Poorly controlled diabetes;
* Recently suffered from hemorrhagic disease or bleeding tendency;
* Recent use of angiotensin-converting enzyme inhibitor (ACEI) drugs;
* Allergic constitution and had a variety of drug allergy history;
* Women in period of pregnancy or lactation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Perfusion Weighted Imaging | 7 days
  Reflect the infarction center and low perfusion of tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurolgy,Xuanwu Hospital of Capital Medical University, Beijing, Beijing Municipality, China